CLINICAL TRIAL: NCT04946487
Title: Effect of the Posterior Ligamentous Complex on the Adjacent Segments Degeneration After Lumbar Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019232
Record Dates: First submitted 2021-06-27; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Adjacent Segment Degeneration; lumbar posterior ligamentous complex; posterior lumbar interbody fusion
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- group 1: patients in this group destructed the posterior ligamentous complex of the adjacent segment
  Interventions: Procedure: total laminectomy
- group 2: patients in this group did not destruct the of the posterior ligamentous complex of the adjacent segment

INTERVENTIONS:
Procedure: total laminectomy — Total laminectomy removes the posterior ligamentous complex (PLC) at the fusion and superior levels.
  Groups: group 1

SUMMARY:
To investigate whether destroying the adjacent posterior ligamentous complex (PLC) has an effect on adjacent segment degeneration (ASD) after L5/S1 posterior lumbar interbody fusion (PLIF)

DETAILED DESCRIPTION:
Purpose: To investigate whether destroying the adjacent posterior ligamentous complex (PLC) has an effect on adjacent segment degeneration (ASD) after L5/S1 posterior lumbar interbody fusion (PLIF).

Methods: This retrospective study was performed in patients who received L5/S1 PLIF with pedicle screw instrumentation for lumbar spinal stenosis with or without isthmic spondylolisthesis. They were divided into the total laminectomy group, which had destruction of the PLC of the adjacent segment, or partial laminectomy group, which did not. Vertebral slip, osteophytes, disk height, and range of motion were examined by plain radiography, and thickness of the ligamentum flavum (LF) and anteroposterior diameters of the lumbar vertebral body and spinal canal were assessed by magnetic resonance imaging (MRI). Disc degeneration and spinal stenosis on MRI scans were categorized. The incidence of ASD and clinical outcome were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* typical clinical symptoms such as disabling low back or leg pain with or without neurological symptoms, intermittent claudication, with refractory to ≥6 months of strict conservative treatment; and L5/S1 single-level PLIF with pedicle screw instrumentation.

Exclusion Criteria:

* previous spine surgery, acute spinal fracture, infection, and tumor.

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From January 2010 to December 2014
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
the Incidences of adjacent segment degeneration | From the end of treatment to more than 8 years
  the Incidences of adjacent segment degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No